CLINICAL TRIAL: NCT01354860
Title: Moxibustion for Knee Osteoarthritis: a Randomized Pilot Clinical Trial
Brief Title: Moxibustion for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Kim, Ki-ok/ President of KIOM, Korea Institute of Oriental Medicine (KIOM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI1002
Record Dates: First submitted 2011-05-04; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-09

CONDITIONS: Idiopathic Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxibustion treatment plus usual care (Experimental)
  Interventions: Other: Moxibustion treatment plus usual care
- usual care alone (No Intervention)
  Interventions: Other: Usual care alone group

INTERVENTIONS:
Other: Moxibustion treatment plus usual care — Treatment group received moxibustion treatment three times a week for 4 consecutive weeks, totally 12 sessions of treatment in addition to usual care to manage their knee OA.
  Moxibustion points include six local acupuncture points on affected knee joint. Up to two additional tender points will be allowed, if necessary. If participants feel knee pain on both knee joints, study practitioners will provide treatment on both knee.
  We will use smokeless indirect moxibustion made of wormwood with a diameter of 1.9 centirmeter and a length of 2.1 centimeter in a cylindrical form for this study (Haitnim Bosung Inc, Korea). Free participant-practitioner interaction will be allowed during the treatment session. Expected total time of each treatment session will be 40 - 60 minutes.
  Other Names: Smokeless indirect moxibustion produced by Haitnim Bosung Inc, Korea.
  Arms: Moxibustion treatment plus usual care
Other: Usual care alone group — Usual care alone group can receive or use any kind of treatment other than moxibustion treatment provided as study intervention, which includes surgery, conventional medication, physical treatment, acupuncture, herbal medicine, over-the-counter drugs and other active treatment. This also applies to the moxibustion treatment group.
  Education material of information on knee osteoarthritis and current management option and self-exercise sheet with a yoga-mat to enhance regular exercise will be provided in both groups at baseline.
  Arms: usual care alone

SUMMARY:
This study aims to assess the feasibility, effectiveness and safety of moxibustion for symptom management and function improvement in patients with knee osteoarthritis, compared to usual care group.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a common joint disease and a leading cause of pain and physical disability in older people. Its symptoms, including pain and physical disability, significantly affect patient's quality of life, and increased depression has been observed in patients with greater pain due to knee OA. Current management options include exercise, weight reduction, Non-steroidal anti-inflammatory drugs (NSAIDs) and other pain medication, intra-articular injections of steroid or hyaluronan, arthroscopic surgery and joint replacement. Except exercise and weight reduction, no known interventions have shown definitive evidence of benefits and safety for knee OA. Thus, it is still worth exploring effective and safe management options for knee OA patients.

Moxibustion is one of traditional Asian medicine using the heat stimulation by burning mugwort (mainly Artemisia vulgaris or Artemisia argyi) on acupuncture points, and regarded as a subtype of acupuncture. Previous literatures reported its use on chronic conditions including gastrointestinal disease, hypertension, musculoskeletal pain, cancer care, gynecological conditions and stroke rehabilitation solely or in combination with routine care or other traditional medicine. However, studies adequately evaluating effects and safety of moxibustion for patients with knee OA are insufficient. Given the gaps between little evidence for effects and safety of moxibustion for knee osteoarthritis and its wide use in clinical practice, the investigators attempted to assess the feasibility, effectiveness and safety of moxibustion for patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 to 70 years old
* Average daily knee pain over 40 points (0-100 point scale)
* diagnosed as knee osteoarthritis according to ACR criteria

Exclusion Criteria:

* Current of past history of inflammatory disease including rheumatoid arthritis
* Cancer
* Traumatic injury which might be related to current knee pain
* Autoimmune disease
* significant deformity of knee joints
* knee replacement surgery on affected knee
* knee arthroscopy within 2 years
* steroid injection in knee joints within 3 months
* viscosupplement injections in knee joints within 6 months
* joint fluid injection within 6 months
* received acupuncture, moxibustion, cupping or herbal medicine within 4 weeks
* uncontrolled hypertension
* diabetes mellitus requiring insulin injection
* life-threatening cardiovascular or neurological events within one year
* chronic respiratory disease
* hemorrhagic disorder
* alcohol or drug addition
* active infectious disease including tuberculosis
* keloidosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
knee pain measured by Western Ontario MacMaster (WOMAC) pain subscale | 4 weeks from baseline
  The primary outcome is the knee pain measured by WOMAC pain subscale at 4 weeks from baseline.

SECONDARY OUTCOMES:
The change from baseline to 4, 8 and 12 weeks in the Short Form Health Survey (SF)-36 | at base line, 4 ,8 and 12 weeks later after allocation
The change from baseline to 4, 8 and 12 weeks in the Beck Depression Inventory(BDI) | at base line, 4 ,8 and 12 weeks later after allocation
The change from baseline to 4, 8 and 12 weeks in the Patient global assessment | 4 ,8 and 12 weeks later after allocation
  Practitioners and participants will evaluate the improvement of knee joint symptoms after treatment. They can chose one of the following 5 grades: Excellent, Good, Fair, Poor and Aggravation.
The change from baseline to 4, 8 and 12 weeks in the physical performance test | at a baseline, 4 ,8 and 12 weeks later after allocation
  Timed-stand test/standing balance test/Six minue walk test
The change from baseline to 4, 8 and 12 weeks in the Numeric Rating Scale (NRS) for pain | at a baseline, 4 ,8 and 12 weeks later after allocation
The change from baseline to 4, 8 and 12 weeks in the Safety measurement | at a baseline, 4 ,8 and 12 weeks later after allocation
The change from baseline to 4, 8 and 12 weeks in the other WOMAC subscale and global score | at base line, 4 ,8 and 12 weeks later after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Sun Mi Choi, PhD, Principal Investigator — Korea Institute of Oriental Medicine
Locations (1):
- Daejeon University Hospital, Daejeon, South Korea